CLINICAL TRIAL: NCT03559595
Title: Increasing Pre-exposure Prophylaxis Among High-Risk African Americans in Louisville KY
Brief Title: Increasing PrEP Among African Americans in Louisville KY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Jelani Kerr, Assistant Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18.0020
Record Dates: First submitted 2018-06-05; First posted 2018-06-18 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: HIV/AIDS PREVENTION

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): All study participants will be exposed to the intervention
  Interventions: Behavioral: Project Prevent

INTERVENTIONS:
Behavioral: Project Prevent — The Project Prevent intervention entails 1) a media campaign to raise PrEP awareness, 2) geographically targeted education initiatives with medical personnel to increase access to consumers, and 3) programming with AIDS service organizations to improve service delivery around PrEP.

SUMMARY:
This study evaluates the effectiveness of a multifaceted strategy to increase pre-exposure prophylaxis (PrEP; a medication regimen to reduce HIV risk) uptake among high risk African Americans in Louisville, KY. We will do this by 1) implementing a media campaign to raise awareness about PrEP, 2) providing PrEP education to medical personnel who can prescribe PrEP, and 3) partnering with AIDS service organizations to improve outreach and linkage to PrEP services.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18-29 years old
* Self-identifies as African American or Black
* Resident of Louisville, KY
* Member of a priority group for PrEP HIV prevention (Men who have sex with men, people who inject drugs, trans women, high risk heterosexuals, people in serodiscordant relationships).
* Not diagnosed with HIV

Exclusion Criteria:

* Older than 29 and younger than 18 years old
* Does not identify as African American or Black
* Does not reside in Louisville, KY
* Not a member of a priority group
* Diagnosed with HIV

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 205 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
PrEP uptake | 12 months
  Reported use of PrEP

SECONDARY OUTCOMES:
PrEP intentions | 12 months
  Intention to use PrEP
PrEP prescription | 12 months
  Prescription of PrEP to eligible individuals by medical personnel

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville, Louisville, Kentucky, United States